CLINICAL TRIAL: NCT01365247
Title: A Randomized Trial of Concurrent Treatment for PTSD and Substance Dependence
Brief Title: Concurrent Treatment for Substance Dependent Individuals With Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Collaborators: Medical University of South Carolina (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Denise Hien, Professor, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DA023187-01A1 (NIH); 1R01DA023187-01A1 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Stress Disorders, Post-Traumatic; Substance-Related Disorders
Keywords: Co-morbid substance disorders and PTSD; Trauma; Alcohol and other drug use disorders; Treatment outcome; Post-Traumatic Stress Disorder (PTSD); Co-morbid Alcohol and other drug use disorders (AOD); Behavioral Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- COPE (Experimental): Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure
  Interventions: Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure
- RPT (Active Comparator): Relapse Prevention Therapy
  Interventions: Behavioral: Relapse Prevention Treatment
- Active Monitoring Control Group (Active Comparator)
  Interventions: Behavioral: Active Monitoring Control Group

INTERVENTIONS:
Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure — A manualized, twelve-week intervention applying cognitive-behavioral strategies and prolonged exposure (PE) techniques to address substance use and trauma related issues.
  Arms: COPE
Behavioral: Relapse Prevention Treatment — Relapse Prevention Treatment is a cognitive-behavioral skills training approach to initiating and maintaining substance use-related goals.
  Arms: RPT
Behavioral: Active Monitoring Control Group — Participants meet with study staff on a weekly basis for the self-monitoring of PTSD and SUD symptoms. Visits consists of self-report assessments, urine toxicology, and a brief check-in with staff to confirm general health and safety.
  Arms: Active Monitoring Control Group

SUMMARY:
This treatment intervention trial is designed for men and women with substance dependence and comorbid Post-Traumatic Stress Disorder (PTSD). Participants will be randomly assigned to one of three conditions (two behavioral treatments [Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure and Relapse Prevention Therapy] and an active monitoring control group) and will be evaluated at baseline and four follow-up points (post-treatment, 1-month, 2- month and 3-month post-treatment).

DETAILED DESCRIPTION:
This study will enhance the knowledge and understanding of concurrently treating individuals with substance use disorders and PTSD in hopes of facilitating treatment retention and increasing the likelihood for more positive treatment outcomes. Following NIDA's stage model for behavior therapies development, this study will take the next step building upon promising findings from Stage IA work with an exposure-based therapy modified to use safely with substance dependent individuals.

This study is a randomized clinical trial to assess the relative efficacy of two active treatment conditions versus an active monitoring control group for substance dependent individuals who also meet criteria for current PTSD according to the diagnostic standards set by the DSM-IV. Eligible participants will be randomly assigned to either: (1) Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE); (2) Relapse Prevention Treatment (RPT) or an (3) Active Monitoring Control Group (AMCG). The study is a three armed randomized controlled trial with repeated outcome measures at post treatment and 1-,2-, and 3-months post-treatment follow-up points for participants in COPE and RPT.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who are a minimum of 18 years and maximum of 65 years.
2. Participants meet DSM-IV criteria for current or past substance dependence
3. Participants must have used alcohol or other drugs within the past 3 months
4. Participants must speak English
5. Participants must meet DSM-IV criteria for current PTSD in response to on an interpersonal, civilian trauma
6. Participants are capable of giving informed consent and capable of complying with study procedures.
7. Participants demonstrate no gross organic mental syndrome

Exclusion Criteria:

1. Participants who are currently suicidal or homicidal
2. Participants who carry a diagnosis of BiPolar I or psychotic disorders are exclusionary.
3. Participants receiving PTSD-specific treatment
4. Participants on anxiolytic, antidepressant or mood stabilizing medications which have been initiated during the 8 weeks prior to study participation
5. Participants refusing to be audio or video taped

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Severity | Six months

SECONDARY OUTCOMES:
Substance Use severity | Six months
Global psychiatric symptom severity | Six months
Treatment retention and compliance | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Hien, Ph.D., Principal Investigator — City College of New York & New York State Psychiatric Institute/Columbia University
Locations (1):
- City College of New York, New York, New York, United States

REFERENCES:
- [Derived] Flanagan JC, Fischer MS, Badour CL, Ornan G, Killeen TK, Back SE. The Role of Relationship Adjustment in an Integrated Individual Treatment for PTSD and Substance Use Disorders Among Veterans: An Exploratory Study. J Dual Diagn. 2017 Jul-Sep;13(3):213-218. doi: 10.1080/15504263.2017.1312039. Epub 2017 May 25. PMID 28541802